CLINICAL TRIAL: NCT01656811
Title: An Efficacy, Safety, and Tolerability Study of Daily Dosing With Levalbuterol, Racemic Albuterol, and Placebo in Pediatric Subjects With Asthma
Brief Title: A Study of Daily Dosing With Levalbuterol, Racemic Albuterol, and Placebo in Pediatric Subjects With Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 051-306
Record Dates: First submitted 2012-07-30; First posted 2012-08-03 (Estimated); Last update posted 2012-08-03 (Estimated); Status verified 2012-07

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Levalbuterol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- levalbuterol 90 mcg (Experimental): levalbuterol 90 mcg delivered via metered dose inhaler (MDI)
  Interventions: Drug: levalbuterol 90 mcg
- levalbuterol 180 mcg (Experimental): levalbuterol 180 mcg delivered via MDI
  Interventions: Drug: levalbuterol 180 mcg
- racemic albuterol 180 mcg (Active Comparator): racemic albuterol 180 mcg delivered via MDI
  Interventions: Drug: racemic albuterol 180 mcg
- Placebo (Placebo Comparator): Placebo delivered via MDI
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: levalbuterol 90 mcg — 90 mcg levalbuterol delivered via MDI 2 actuations of 45 mcg QID
  Arms: levalbuterol 90 mcg
Drug: levalbuterol 180 mcg — 180 mcg levalbuterol delivered via MDI 2 actuations of 90 mcg QID
  Arms: levalbuterol 180 mcg
Drug: racemic albuterol 180 mcg — 180 mcg racemic albuterol delivered via MDI 2 actuations of 90 mcg QID
  Arms: racemic albuterol 180 mcg
Drug: Placebo — Placebo 2 actuations QID
  Arms: Placebo

SUMMARY:
Multicenter, randomized, double-blind, placebo- and active-controlled, Phase II, parallel-group study of up to four weeks in duration. The study consisted of a screening visit followed by a one-week single blind placebo period. At next visit, each subject was randomized to one of four treatment groups: 90 mcg levalbuterol, 180 mcg levalbuterol, 180 mcg racemic albuterol, or placebo. All study medication was administered as 2 actuations 4 times a day for 21 days.

DETAILED DESCRIPTION:
This was a multicenter, randomized, double-blind, placebo- and active-controlled, Phase II, parallel-group study up to four weeks in duration. Seven days of QID (four times a day) single-blind, placebo administration (via metered dose inhaler (MDI)) was followed by 21 days of QID double-blind treatment. During the single-blind period, rescue medication consisted of racemic albuterol MDI (90 mcg per actuation) for all subjects. During the double-blind period, rescue medication consisted of double-blind levalbuterol MDI (45 mcg per actuation) for all subjects in the levalbuterol treatment groups or double-blind racemic albuterol MDI (90 mcg per actuation) for all subjects in the racemic albuterol and placebo treatment groups.The study consisted of two periods, an optional follow-up visit, and a final telephone evaluation. This study was previously conducted by Sepracor Inc. In October 2009, Sepracor Inc. was acquired by Dainippon Sumitomo Pharma., and in October 2010, Sepracor Inc's name was changed to Sunovion Pharmaceuticals Inc.

ELIGIBILITY:
Inclusion Criteria:

* Subject's parent/legal guardian provided written informed consent prior to participation in the study.
* Subject and the subject's parent/legal guardian were willing and able to comply with the study procedures and visit schedules.
* Subject (male or female) was between the ages of 4 to 11 years (inclusive) at the time of consent.
* Female subject 8 years of age or older had a negative serum pregnancy test at screening.
* Subject had a documented diagnosis of asthma for a minimum of 6 months prior to screening, as defined by the AARC.
* Subject demonstrated a baseline FEV1 within greater than or equal to 45% and less than or equal to 80% of predicted for their height, age, gender, and race
* Following abstention from medications used to treat asthma subject demonstrated greater than or equal to 12% reversibility of airflow obstruction within 15-30 minutes following inhalation of 180 mcg (2 actuations of 90 mcg) racemic albuterol MDI.
* Subject had stable baseline asthma (in the opinion of the Investigator) and had been using a beta-adrenergic agonist and/or anti-asthma anti-inflammatory medication, and/or over-the-counter asthma medication for at least 6 months prior to screening.
* Subject was in good health (with the exception of asthma) and not suffering from any chronic condition that might affect their respiratory function.
* Subject had a chest x-ray that was not diagnostic of pneumonia, atelectasis, pulmonary fibrotic disease, pneumothorax, chronic obstructive pulmonary disease, etc. The most recent chest x-ray taken within 12 months prior to randomization was allowed to be used.
* Subject's parent/legal guardian was able to complete diary cards and medical event calendars reliably on a daily basis, understand dosing instructions and questionnaire completion, and demonstrate how to use the MiniWright PEF meter to complete morning and evening peak expiratory flow measurements.

Exclusion Criteria:

* Subject was expected to require parenteral corticosteroids, adrenergic bronchodilators, non-prescription asthma medications, or ipratropium bromide as per list below:

Corticosteroids - Parenteral = 30 days wash out period. Adrenergic bronchodilators - Inhaled, short-acting = greater than or equal to 7 hours wash out period, Nebulized, short acting = greater than or equal to 10 hours wash out period, Inhaled, long acting = greater than or equal to 24 hours wash out period, Oral QID or TID preparation =greater than or equal to 24 hours wash out period, Oral BID preparations = greater than or equal to 36 hours wash out period, Nonprescription asthma medications = greater than or equal to 48 hours wash out period, Ipratropium bromide = greater than or equal to 48 hours wash out period (Study medication and rescue medication were allowed to be used as needed but were required to be with-held prior to Study visits according to the schedule noted above)

* Female subject was pregnant or lactating.
* Subject participated in an investigational drug study within 30 days prior to screening, or was currently participating in another clinical trial.
* Subject had a schedule that prevented him or her from taking the first daily dose of study medication and/or starting study visits before 9 AM.
* Subject had travel commitments during the study that would have interfered with trial measurements and/or compliance.
* Subject had a history of hospitalization for asthma within 60 days prior to screening, or was scheduled for in-patient hospitalization, including elective surgery during the course of the trial.
* Subject had a known sensitivity to levalbuterol or racemic albuterol, including Ventolin or any of the excipients contained in any of these formulations.
* Subject was using any prescription drug with which albuterol sulfate administration was contraindicated
* Subject was currently diagnosed with life-threatening asthma, defined as a history of asthma episodes requiring intubation, associated with hypercapnia, respiratory arrest, or hypoxic seizures within 12 months prior to screening..
* Subject had clinically significant abnormalities that may have interfered with the metabolism or excretion of the study drug (e.g., abnormalities of the renal, hepatic, metabolic, or endocrine function).
* Subject had a history of cancer.
* Subject had hyperthyroidism, diabetes, hypertension, cardiac diseases, or seizure disorders that were not well controlled by medication or that may have interfered with the successful completion of this protocol.
* Subject had a history of substance abuse or drug abuse within 12 months prior to screening.
* Subject had a documented history of bronchopulmonary aspergillosis or any form of allergic alveolitis.
* Subject suffered from a clinically significant upper or lower respiratory tract infection in the 2 weeks prior to screening. (Note: Any subject who developed a clinically significant respiratory tract infection during the study was required to be discontinued.)
* Subject had clinically significant abnormal laboratory values (hematology, blood chemistry, or urinalysis).
* Subject had a clinically significant abnormal 12-lead ECG that would have put the subject at risk for experiencing adverse cardiac events.
* Subject had a history of cigarette smoking or use of other tobacco products.
* Subject was a staff member or a relative of a staff member at the time of the study.

Ages: 4 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 146 (Actual)
Dates: Start 2001-10; Primary Completion 2002-07 (Actual); Study Completion 2002-07 (Actual)

PRIMARY OUTCOMES:
Peak percent change in FEV1 (forced expiratory volume in one second) from visit predose averaged over the double-blind period to investigate the efficacy of levalbuterol versus racemic albuterol | Week 0-4

SECONDARY OUTCOMES:
Plasma concentrations of (R)-albuterol and (S)-albuterol over time to determine the pharmacokinetics of levalbuterol in pediatric subjects with asthma | Week 0-4
Number of AEs to compare the safety and tolerability of two different doses of levalbuterol | Week 0-4

CONTACTS AND LOCATIONS:
Overall Officials: Xopenex Medical Director, MD, Study Director — Sumitomo Pharma America, Inc.